CLINICAL TRIAL: NCT01210560
Title: A Multi-center, Parallel-group, Randomized, Double-blind, Placebo-masked, Multiple Dose Trial of Modified-release (MR) and Immediate-release (IR) Tolvaptan in Subjects With Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Brief Title: Dose-finding Study of New Tolvaptan Formulation in Subjects With ADPKD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 156-09-285
Record Dates: First submitted 2010-09-21; First posted 2010-09-28 (Estimated); Results first posted 2018-06-14 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-05

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
Keywords: Kidney Disease; Polycystic Kidney Disease
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Kidney Diseases; Polycystic Kidney Diseases | interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 20 mg MR (Experimental)
  Interventions: Drug: Tolvaptan MR
- 40 mg MR (Experimental)
  Interventions: Drug: Tolvaptan MR
- 60 mg MR (Experimental)
  Interventions: Drug: Tolvaptan MR
- 120 mg MR (Experimental)
  Interventions: Drug: Tolvaptan MR
- 120 mg IR (Experimental)
  Interventions: Drug: Tolvaptan IR

INTERVENTIONS:
Drug: Tolvaptan MR — 20 mg Tolvaptan MR capsule(morning); Placebo capsules/tablets (morning and afternoon) for 7 days
  Other Names: OPC-41061
  Arms: 20 mg MR
Drug: Tolvaptan MR — 20 mg Tolvaptan MR capsule(morning and afternoon); Placebo capsules/tablets (morning and afternoon) for 7 days
  Other Names: OPC-41061
  Arms: 40 mg MR
Drug: Tolvaptan MR — 60 mg Tolvaptan MR capsule(morning); Placebo capsules/tablets (morning and afternoon) for 7 days
  Other Names: OPC-41061
  Arms: 60 mg MR
Drug: Tolvaptan IR — 90 mg Tolvaptan IR tablet(morning); 30 mg Tolvaptan IR tablet (afternoon); Placebo capsules (morning and afternoon) for 7 days
  Other Names: OPC-41061
  Arms: 120 mg IR
Drug: Tolvaptan MR — 120 mg Tolvaptan MR capsule(morning); Placebo capsules/tablets (morning and afternoon) for 7 days
  Other Names: OPC-41061
  Arms: 120 mg MR

SUMMARY:
To establish pharmacokinetics (PK), pharmacodynamics (PD), and adverse event (AE) profile of tolvaptan administered as the modified-release (MR) formulation in ADPKD subjects. The goals of this trial are two-fold:

1. To directly compare the immediate release (IR) and MR formulations
2. To determine the dose range and dose regimen for MR (dose finding)

DETAILED DESCRIPTION:
Group 1 will have 12 subjects enrolled in a 3-period, randomized, crossover to compare multiple doses of a 90-30 mg split-dose of the tolvaptan IR formulation, a 120 mg once daily (QD) dose of the tolvaptan MR formulation, and, in an incomplete block randomization, multiple doses of either 20 mg QD, 60 mg QD, or 20 mg twice daily (BID) tolvaptan MR formulation. All dose regimens will be administered for 7 days. Placebo doses will be administered in order to mask QD vs BID treatments.

Group 2 will have 12 subjects enrolled in a 3-period, randomized, crossover to compare multiple oral doses of the tolvaptan MR formulation administered for 7 days as 20 mg QD, 60 mg QD, and 20 mg BID. Placebo capsules will be administered in order to mask QD vs BID treatments.

Subjects will have in-clinic assessments on 12 days to obtain 24-hour PK and PD data. Subjects will visit the clinic from the afternoon of Day -1 through the morning of Day 1. They will return at the end of each dosing period for a similar inpatient period (ie, from the afternoon of Day 6 through the morning of Day 8, from the afternoon of Day 13 through the morning of Day 15, from the afternoon of Day 20 through the morning of Day 22). Except for the first dose of each period and the doses taken in the clinic on the last day of each regimen and the afternoon of Days 6, 13 and 20, all other doses will be taken by the subject as an outpatient.

ELIGIBILITY:
Inclusion Criteria:

* Subjects (male or female) who are surgically sterile (ie, have undergone hysterectomy) or using contraception or agree to remain abstinent
* Subjects between the ages of 18 and 50, inclusive
* Subjects with a body mass index between 19 to 35 kg/m2 (inclusive)
* Subjects with a diagnosis of ADPKD by modified Ravine criteria
* Subjects must be in good health as determined by medical history, physical examination, ECG, serum/urine biochemistry, hematology, and serology tests
* Subjects with the ability to provide written, informed consent prior to initiation of any trial-related procedures, and ability, in the opinion of the principle investigator, to comply with all requirements of the trial
* Subjects who expect to be able to complete all dosing periods and assessments within 42 (+2) days after dosing on Day 1

Exclusion Criteria:

* Subjects using diuretics within 14 days prior to check in on Day -1
* Subjects with incontinence, overactive bladder, or urinary retention (eg, benign prostatic hyperplasia)
* Subjects (male or female) with nocturia/urgency (outside of the 2 to 4 times awakening per night expected for ADPKD patients) at screening
* Subjects with liver disease, liver function abnormalities or serology other than that expected for ADPKD with cystic liver disease at baseline
* Subjects with clinically significant abnormality in past medical history, or at the Screening physical examination, that in the investigator's or sponsor's opinion may place the volunteer at risk or interfere with outcome variables including absorption, distribution, metabolism, and excretion of drug. This includes, but is not limited to, history of or concurrent cardiac, hepatic, renal, neurologic, endocrine, gastrointestinal, respiratory, hematologic, and immunologic disease
* Subjects with a history of drug and/or alcohol abuse within 2 years prior to screening
* Subjects who have a history of or test positive at screening for hepatitis B surface antigen (HBsAg), hepatitis C antibodies (anti-HCV), and/or human immunodeficiency virus (HIV)
* Subjects who have clinically significant allergic reactions to tolvaptan or chemically related structures such as benzazepines (eg, benzazepril, conivaptan, fenoldopam mesylate or mirtazapine)
* Subjects who have taken an investigational drug within 30 days preceding trial entry
* Subjects with any history of significant bleeding or hemorrhagic tendencies
* Subjects with a history of difficulty in donating blood
* Subjects who have donated blood or plasma within 30 days prior to dosing
* Subjects who have consumed alcohol and/or food or beverages containing methylxanthines, grapefruit, grapefruit juice, Seville oranges, or Seville orange juice within 72 hours prior to Day 1 dosing
* Subjects taking CYP3A4 inhibitors, with the exception of amiodarone, taken within 30 days of dosing (eg, amprenavir, atorvastatin, aprepitant, chloramphenicol [not eye drops], cimetidine, clarithromycin, clotrimazole [if used orally], danazol, delavirdine, diltiazem, erythromycin, fluconazole, fluvoxamine, indinavir, isoniazid, itraconazole, josamycin, ketoconazole, nelfinavir, nefazadone, quinupristin/dalfopristin, ritonavir, saquinavir, troleandomycin, verapamil)
* Subjects taking CYP3A4 inducers taken within 7 days of dosing (eg, rifampin, St. Johns Wort)
* Subjects with a history of serious mental disorders
* Subjects with previous exposure to tolvaptan

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2010-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Czerwiec, M.D., Ph.D., Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (6):
- United States (6):
  - Tufts-New England Medical Center, Boston, Massachusetts
  - Davita Clinical Research, Minneapolis, Minnesota
  - Mayo Medical Center, Rochester, Minnesota
  - University Hospitals of Cleveland/Case, Cleveland, Ohio
  - Northwest Renal Clinic Inc., Portland, Oregon
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039
- [Derived] Gobburu J, Ivaturi V, Wang X, Shoaf SE, Jadhav P, Perrone RD. Comparing Effects of Tolvaptan and Instruction to Increase Water Consumption in ADPKD: Post Hoc Analysis of TEMPO 3:4. Kidney360. 2023 Dec 1;4(12):1702-1707. doi: 10.34067/KID.0000000000000302. Epub 2023 Nov 21. PMID 37986188

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 6 centers in the United States. 25 participants were randomized (12+13) to Group 1 & 2 with 5 & 3 treatment sequences, respectively; received tolvaptan Modified-release [MR] capsules & Immediate-release [IR] tablets in Group 1 & MR in Group 2 over 3 therapy periods (each 7 days) in parallel-group, crossover design
Pre-assignment Details: Screening visit, baseline visit, 3 periods - each with 3 treatments in Group 1 & 2 in one of the sequences DAE, DBE, DCE, EAD, EBD / ECD & FGH, HFG / GHF (2 & 4 participants per sequence) respectively; (MR: A&F= 20mg, B&G = 20+20mg, C&H = 60mg, D = 120mg; IR: E = 90+30mg) and 7 Day follow-up. All doses were taken orally once/twice(B&G) daily.
Groups:
- Group 1: DAE: D = participants received MR tolvaptan 120 mg QD A = participants received MR tolvaptan 20 mg QD E = participants received IR tolvaptan 90 + 30 mg QD
- Group 1: DBE: D = participants received MR tolvaptan 120 mg QD B = participants received MR tolvaptan 20 mg BID E = participants received IR tolvaptan 90 + 30 mg QD
- Group 1: DCE: D = participants received MR tolvaptan 120 mg QD C = participants received MR tolvaptan 60 mg QD E = participants received IR tolvaptan 90 + 30 mg QD
- Group 1: EAD: E = participants received IR tolvaptan 90 + 30 mg QD A = participants received MR tolvaptan 20 mg QD D = participants received MR tolvaptan 120 mg QD
- Group 1: EBD: E = participants received IR tolvaptan 90 + 30 mg QD B = participants received MR tolvaptan 20 mg BID D = participants received MR tolvaptan 120 mg QD
- Group 1: ECD: E = participants received IR tolvaptan 90 + 30 mg QD C = participants received MR tolvaptan 60 mg QD D = participants received MR tolvaptan 120 mg QD
- Group 2: FGH: F = participants received MR tolvaptan 20 mg QD G = participants received MR tolvaptan 20 + 20 mg BID H = participants received MR tolvaptan 60 mg QD
- Group 2: HFG: H = participants received MR tolvaptan 60 mg QD F = participants received MR tolvaptan 20 mg QD G = participants received MR tolvaptan 20 + 20 mg BID
- Group 2: GHF: G = participants received MR tolvaptan 20 + 20 mg BID H = participants received MR tolvaptan 60 mg QD F = participants received MR tolvaptan 20 mg QD
Period: Intervention 1 (7 Days)
Arm/Group | Group 1: DAE | Group 1: DBE | Group 1: DCE | Group 1: EAD | Group 1: EBD | Group 1: ECD | Group 2: FGH | Group 2: HFG | Group 2: GHF
Started | 2 | 2 | 2 | 2 | 2 | 2 | 4 | 4 | 5
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 4 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Intervention 2 (7 Days)
Arm/Group | Group 1: DAE | Group 1: DBE | Group 1: DCE | Group 1: EAD | Group 1: EBD | Group 1: ECD | Group 2: FGH | Group 2: HFG | Group 2: GHF
Started | 2 | 2 | 2 | 2 | 2 | 2 | 4 | 4 | 5
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 4 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Intervention 3 (7 Days)
Arm/Group | Group 1: DAE | Group 1: DBE | Group 1: DCE | Group 1: EAD | Group 1: EBD | Group 1: ECD | Group 2: FGH | Group 2: HFG | Group 2: GHF
Started | 2 | 2 | 2 | 2 | 2 | 2 | 4 | 4 | 5
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 4 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Group 1 participants enrolled in a 3-period, randomized, crossover design to compare multiple doses of a 90+30 mg split-dose of the tolvaptan IR formulation, a 120 mg QD dose of the tolvaptan MR formulation, and, in an incomplete block randomization, multiple doses of either 20 mg QD, 60 mg QD, or 20 mg BID tolvaptan MR formulation. All dose regimens were administered for 7 days. Placebo doses were administered in order to mask formulation and dosing regimen.
- Group 2: Group 2 participants enrolled in a 3-period, randomized, crossover design to compare multiple oral doses of the tolvaptan MR formulation administered for 7 days as 20 mg QD, 60 mg QD, and 20 mg BID. Placebo capsules were administered in order to mask dosing regimen.
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.4 (4.3) | 36.8 (9.0) | 38.0 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 5 | 9 | 14

OUTCOME MEASURES:

1. Primary Outcome: Maximum (Peak) Plasma Concentration of the Drug [Cmax] and Minimum (Trough) Plasma Concentration of the Drug [Cmin] After Tolvaptan Treatment on Day 7.
Description: Blood samples (6 mL) for determination of tolvaptan PK parameters were collected on Day 1 predose, and on Days 7, 14 and 21 at predose, and 1, 2, 4, 6, 8, 9, 10, 12, 16, and 24 hours postdose. If a sample was not drawn at the designated time, a window of ± 3 minutes for each blood draw was acceptable. Maximum and minimum plasma concentration of the drug was calculated.
Time Frame: Day 7
Population: Participants having valid measurements (per clinical pharmacology) were included.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- MR 20 mg: Participants received MR tolvaptan 20 mg QD.
- MR 20+20 mg: Participants received MR tolvaptan 20 mg BID.
- MR 60 mg: Participants received MR tolvaptan 60 mg QD.
- MR 120 mg: Participants received MR tolvaptan 120 mg QD.
- IR 90+30 mg: Participants received IR tolvaptan 90+30 mg QD.
Arm/Group | MR 20 mg | MR 20+20 mg | MR 60 mg | MR 120 mg | IR 90+30 mg
Number analyzed (Participants) | 17 | 16 | 17 | 12 | 12
ng/mL
  Cmax | 140 (68.4) | 175 (60.1) | 350 (156) | 669 (370) | 716 (344)
  Cmin | 14.7 (9.95) | 50.8 (24.0) | 51.1 (32.3) | 139 (75.5) | 57.5 (41.8)

2. Primary Outcome: Time to Maximum (Peak) Plasma Concentration (Tmax) After Tolvaptan Treatment on Day 7.
Description: Blood samples (6 mL) for determination of tolvaptan PK parameters were collected on Day 1 predose, and on Days 7, 14 and 21 at predose, and 1, 2, 4, 6, 8, 9, 10, 12, 16, and 24 hours postdose. If a sample was not drawn at the designated time, a window of ± 3 minutes for each blood draw was acceptable. Time to maximum plasma concentration was calculated.
Time Frame: Day 7
Population: Participants having valid measurements (per clinical pharmacology) were included.
Measure: Median (Full Range); unit: Hours
Arm/Group | MR 20 mg | MR 20+20 mg | MR 60 mg | MR 120 mg | IR 90+30 mg
Number analyzed (Participants) | 17 | 16 | 17 | 12 | 12
Hours | 6.00 [3.97 to 10.00] | 6.00 [3.97 to 16.00] | 6.00 [3.98 to 9.00] | 5.98 [3.97 to 6.00] | 2.00 [1.00 to 9.00]

3. Primary Outcome: Area Under the Concentration-time Curve During the Dosing Interval at Steady State and Area Under the Concentration-time Curve From Time 0 to 24 Hours Postdose (AUCT & AUC0-24h) After Tolvaptan Treatment on Day 7.
Description: Blood samples (6 mL) for determination of tolvaptan PK parameters were collected on Day 1 predose, and on Days 7, 14 and 21 at predose, and 1, 2, 4, 6, 8, 9, 10, 12, 16, and 24 hours postdose. If a sample was not drawn at the designated time, a window of ± 3 minutes for each blood draw was acceptable. Hence, both AUCT and AUC0-24h values were calculated.
Time Frame: Day 7
Population: Participants having valid measurements (per clinical pharmacology) were included.
Measure: Mean (Standard Deviation); unit: ng·h/mL
Arm/Group | MR 20 mg | MR 20+20 mg | MR 60 mg | MR 120 mg | IR 90+30 mg
Number analyzed (Participants) | 17 | 16 | 17 | 12 | 12
ng·h/mL | 1260 (654) | 2310 (704) | 3600 (1670) | 7740 (3650) | 6570 (3230)

4. Secondary Outcome: Number of Participants With Urine Osmolality < 300 mOsm/kg at 23.5 Hours Postdose.
Description: For determination of duration of urine osmolality <300 mOsm/kg, the value was the end time of the last collection interval in which urine osmolality was <300 mOsm/kg. Day 8 in the table below was defined as Day 8 of Period 1, Day 15 of Period 2, and Day 22 of period 3.
Time Frame: 23.5 hours post-dose
Population: All participants who had taken study drug and had measurements of the pharmacodynamic endpoint were included.
Measure: Count of Participants; unit: Participants
Arm/Group | MR 20 mg | MR 20+20 mg | MR 60 mg | MR 120 mg | IR 90+30 mg
Number analyzed (Participants) | 17 | 17 | 17 | 12 | 12
Participants
  Baseline | 1 | 1 | 1 | 0 | 0
  Day 8: number analyzed (Participants) | 17 | 16 | 16 | 12 | 12
  Day 8 | 5 | 11 | 9 | 11 | 11

5. Secondary Outcome: Change From Baseline in Urine Osmolality Area Under the Concentration-time Curve From Time 0 to 24 Hours Postdose (AUC0-24h) at Day 7.
Description: The AUC0-24h for urine osmolality was determined by multiplying the concentration by the collection interval duration for each collection interval and summing all the intervals in the 24-hour period. If the urine volume for an interval is zero, the duration of that interval will be added to the next collection interval. Day 7 was defined as Day 7 of Period 1, Day 14 of Period 2 and Day 21 of Period 3.
Time Frame: Day 7
Population: All participants who had taken study drug and had measurements of the pharmacodynamic endpoint were included.
Measure: Mean (Standard Deviation); unit: mOsm/kg*Hour
Arm/Group | MR 20 mg | MR 20+20 mg | MR 60 mg | MR 120 mg | IR 90+30 mg
Number analyzed (Participants) | 17 | 16 | 17 | 12 | 11
mOsm/kg*Hour | -2546 (1743) | -3438 (2277) | -4209 (2569) | -4325 (2237) | -4620 (2419)

6. Secondary Outcome: Change From Baseline in Urine Osmolality at Day 7.
Description: To determine the tolerability and nighttime urinary suppression of osmolality. The urine osmolality was summarized by collection interval (0 to 4, 4 to 8, 8 to 12, 12 to 16, and 16 to 24 hours)
Time Frame: 0-4, 4-8, 8-12, 12-16, 16-24 Hours at Day 7
Population: All participants who had taken study drug and have measurements of the pharmacodynamic endpoint were included.
Measure: Mean (Standard Deviation); unit: mOsm/kg
Arm/Group | MR 20 mg | MR 20+20 mg | MR 60 mg | MR 120 mg | IR 90+30 mg
Number analyzed (Participants) | 17 | 17 | 17 | 12 | 12
mOsm/kg
  0-4 Hour: number analyzed (Participants) | 17 | 16 | 17 | 12 | 12
  0-4 Hour | 2.6 (132.1) | -0.7 (111.9) | -88.9 (130.9) | -59.5 (169.2) | -123.3 (139.5)
  4-8 Hour: number analyzed (Participants) | 17 | 16 | 17 | 12 | 12
  4-8 Hour | -140.9 (127.1) | -128.3 (127.2) | -188.2 (140.5) | -186.1 (161.1) | -191.8 (155.1)
  8-12 Hour: number analyzed (Participants) | 17 | 16 | 17 | 12 | 12
  8-12 Hour | -123.1 (115.9) | -172.1 (129.8) | -201.8 (158.8) | -167.1 (148.7) | -166.9 (131.7)
  12-16 Hour: number analyzed (Participants) | 17 | 16 | 17 | 12 | 11
  12-16 Hour | -128.3 (142.9) | -193.6 (152.5) | -195.8 (151.6) | -176.3 (121.8) | -178.3 (128.9)
  16-24 Hour: number analyzed (Participants) | 17 | 16 | 17 | 12 | 12
  16-24 Hour | -123.4 (102.6) | -182.4 (145.6) | -188.8 (160.0) | -246.1 (108.9) | -239.8 (117.8)

7. Secondary Outcome: Change From Baseline in Urine Volume at 24 Hours at Day 7.
Description: Urine volume was collected by 0 to 24-hour interval at Day 7. Day 7 was defined as Day 7 of Period 1, Day 14 of Period 2 and Day 21 of Period 3.
Time Frame: Day 7
Population: All participants who had taken study drug and have measurements of the pharmacodynamic endpoint were included.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | MR 20 mg | MR 20+20 mg | MR 60 mg | MR 120 mg | IR 90+30 mg
Number analyzed (Participants) | 17 | 16 | 16 | 12 | 12
mL | 1111 (919) | 2066 (1237) | 2396 (1022) | 3722 (1776) | 3820 (1759)

8. Secondary Outcome: Change From Baseline in Urine Volume by Interval at Day 7.
Description: Urine volume collected was by interval (0-4, 4-8, 8-12, 12-16, 16-24 hours). Day 7 was defined as Day 7 of Period 1, Day 14 of Period 2 and Day 21 of Period 3.
Time Frame: 0-4, 4-8, 8-12, 12-16, 16-24 Hours at Day 7
Population: All participants who had taken study drug and have measurements of the pharmacodynamic endpoint were included.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | MR 20 mg | MR 20+20 mg | MR 60 mg | MR 120 mg | IR 90+30 mg
Number analyzed (Participants) | 17 | 17 | 17 | 12 | 12
mL
  0-4 Hour: number analyzed (Participants) | 17 | 16 | 17 | 12 | 12
  0-4 Hour | -87 (348) | -118 (391) | 56 (345) | 87 (449) | 241 (412)
  4-8 Hour: number analyzed (Participants) | 17 | 16 | 17 | 12 | 12
  4-8 Hour | 326 (531) | 423 (439) | 636 (382) | 785 (605) | 825 (472)
  8-12 Hour: number analyzed (Participants) | 17 | 16 | 17 | 12 | 12
  8-12 Hour | 301 (317) | 529 (349) | 689 (603) | 887 (558) | 801 (494)
  12-16 Hour: number analyzed (Participants) | 17 | 16 | 16 | 12 | 12
  12-16 Hour | 314 (328) | 635 (473) | 667 (337) | 926 (459) | 910 (738)
  16-24 Hour: number analyzed (Participants) | 17 | 16 | 17 | 12 | 12
  16-24 Hour | 257 (407) | 598 (482) | 286 (421) | 1038 (642) | 1044 (421)

9. Secondary Outcome: Duration of Urine Osmolality Less Than 300 mOsm/kg at Baseline and Day 7.
Description: Duration of urine osmolality remains below 300 mOsm/kg was the sum of the durations (nominal times) of all intervals where the urine concentration was < 300 mOsm/kg. Day 7 was defined as Day 7 of Period 1, Day 14 of Period 2, and Day 21 of Period 3.
Time Frame: Baseline and Day 7
Population: The duration that urine osmolality remained < 300 mOsm/kg was not calculated. Instead was calculated as the sum where urine osmolality was < 300 mOsm/kg in the 24-hour postdose period. The change was made because low doses of the MR formulation frequently do not produce suppression of urine osmolality in the 0- to 4-hour period.
Measure: Median (Full Range); unit: Hours
Arm/Group | MR 20 mg | MR 20+20 mg | MR 60 mg | MR 120 mg | IR 90+30 mg
Number analyzed (Participants) | 17 | 17 | 17 | 12 | 12
Hours
  Baseline | 8.0 [0 to 24.0] | 8.0 [0 to 24.0] | 8.0 [0 to 24.0] | 14.0 [0 to 24.0] | 14.0 [0 to 24.0]
  Day 7: number analyzed (Participants) | 17 | 16 | 17 | 12 | 12
  Day 7 | 16.0 [4.0 to 24.0] | 24.0 [4.0 to 24.0] | 24.0 [8.0 to 24.0] | 24.0 [20.0 to 24.0] | 24.0 [24.0 to 24.0]

10. Secondary Outcome: Change From Baseline in Number of Urine Voids During Awake Periods.
Description: Average number of daily urine voids during awake periods for each dose group. Day 1 was defined as Day1 of Period 1, Day 8 of Period 2 adn Day 15 of Period 3; Day 7 was defined as Day 7 of Period 1, Day 14 of Period 2 and Day 21 of Period 3; Same rule applied to Day 2 and Day 6.
Time Frame: Days 1, 2, 3, 4, 5, 6 and 7
Population: All participants who had taken study drug and had measurements of the pharmacodynamic endpoint were included.
Measure: Mean (Standard Deviation); unit: Number of urine voids
Arm/Group | MR 20 mg | MR 20+20 mg | MR 60 mg | MR 120 mg | IR 90+30 mg
Number analyzed (Participants) | 17 | 17 | 17 | 12 | 12
Number of urine voids
  Day 1 | 1.7 (4.1) | 1.5 (3.1) | 3.5 (4.3) | 5.6 (5.6) | 4.8 (4.1)
  Day 2 | -0.4 (2.9) | 1.2 (4.0) | 1.8 (4.1) | 4.8 (7.8) | 3.8 (4.2)
  Day 3 | -0.8 (2.4) | 0.9 (2.4) | 2.4 (3.9) | 3.1 (4.6) | 3.3 (5.2)
  Day 4 | -1.4 (2.3) | 1.5 (3.8) | 0.4 (5.0) | 2.8 (5.0) | 3.7 (5.9)
  Day 5 | -0.5 (2.9) | 0.6 (3.5) | -0.4 (4.2) | 3.3 (5.6) | 4.0 (4.9)
  Day 6 | 0.0 (3.3) | 2.9 (4.1) | 5.8 (10.6) | 2.3 (6.8) | 4.8 (5.2)
  Day 7: number analyzed (Participants) | 17 | 16 | 17 | 12 | 12
  Day 7 | 2.0 (3.0) | 3.5 (2.4) | 3.5 (3.8) | 2.8 (6.4) | 4.3 (4.5)

11. Secondary Outcome: Change From Baseline in Number of Urine Voids During Sleep Periods.
Description: Average number of daily urine voids during sleep periods for each dose group. Day 1 was defined as Day 1 of Period 1, Day 8 of Period 2, Day 15 of Period 3; Day 7 was defined as Day 7 of Period 1, Day 14 of Period 2 and Day 21 of Period 3; Same rule applied to Day 2 to 6.
Time Frame: Days 1, 2, 3, 4, 5, 6 and 7
Population: All participants who had taken study drug and have measurements of the pharmacodynamic endpoint were included.
Measure: Mean (Standard Deviation); unit: Number of urine voids
Groups:
- MR 60 mg: Participants received MR tolvaptan 60 mg Q
Arm/Group | MR 20 mg | MR 20+20 mg | MR 60 mg | MR 120 mg | IR 90+30 mg
Number analyzed (Participants) | 17 | 17 | 17 | 12 | 12
Number of urine voids
  Day 1 | 0.6 (1.6) | 1.1 (2.0) | 0.4 (2.2) | 2.5 (1.7) | 1.5 (1.6)
  Day 2 | -0.2 (1.7) | 0.8 (1.6) | 0.8 (1.9) | 1.8 (1.4) | 1.7 (1.2)
  Day 3 | 0.1 (1.0) | 1.4 (2.4) | 0.8 (1.7) | 1.9 (1.5) | 1.9 (1.7)
  Day 4 | 0.6 (2.3) | 0.7 (1.6) | 0.5 (1.7) | 1.7 (1.3) | 1.8 (1.9)
  Day 5 | 0.3 (1.3) | 0.9 (2.0) | 0.2 (1.4) | 1.0 (2.0) | 0.9 (1.7)
  Day 6 | 1.2 (3.3) | 1.3 (2.0) | 0.4 (1.6) | 1.1 (2.1) | 1.7 (1.7)
  Day 7: number analyzed (Participants) | 17 | 16 | 17 | 12 | 12
  Day 7 | 0.1 (1.3) | 1.0 (1.7) | 0.9 (1.8) | 1.8 (2.4) | 2.1 (1.9)

12. Secondary Outcome: Change From Baseline in Symptom Burden by Autosomal Dominant Polycystic Kidney Disease (ADPKD) Nocturia Quality of Life Questionnaire at Day 6.
Description: In ADPKD Nocturia Quality of Life Questionnaire, questions 1 to 11 (with possible scores ranging from 0 to 4 and higher scores indicating better quality of life) were pooled to provide a total score (maximum of 44 points). Response scores of Question 12 (with possible scores ranging from 1 to 10, with higher scores indicating more interference (worse quality of life) with everyday life due to urination at night) were pooled separately. Day 6 was defined as Day 6 of Period 1, Day 13 of Period 2 and Day 20 of Period 3.
Time Frame: Day 6
Population: All participants who had taken study drug and have measurements of the pharmacodynamic endpoint were included.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | MR 20 mg | MR 20+20 mg | MR 60 mg | MR 120 mg | IR 90+30 mg
Number analyzed (Participants) | 17 | 17 | 17 | 12 | 12
Units on a scale
  Nocturia Quality of life Question (Q) 1 To Q 11 | -1.5 (4.3) | -6.9 (9.9) | -5.1 (7.6) | -15.0 (13.3) | -13.1 (12.3)
  Nocturia Quality of life Q 12 | 0.6 (1.3) | 1.9 (2.7) | 1.4 (2.5) | 4.2 (3.6) | 3.7 (3.5)

13. Secondary Outcome: Number of Participants Experiencing Urinary Urgency Based on Urinary Urgency Questionnaire (Question 1) at Baseline and Day 6.
Description: For the ADPKD Urinary Urgency Questionnaire, Question 1 (currently experiencing urgency?) was assigned 'Yes' or 'No' to measure current urine urgency status. Baseline was defined as last pre-dose evaluation; Day 6 was defined as Day 6 of Period 1, Day 13 of Period 2 and Day 20 of Period 3.
Time Frame: Baseline and Day 6
Population: All participants who had taken study drug and have measurements of the pharmacodynamic endpoint were included.
Measure: Number; unit: Participants
Arm/Group | MR 20 mg | MR 20+20 mg | MR 60 mg | MR 120 mg | IR 90+30 mg
Number analyzed (Participants) | 17 | 17 | 17 | 12 | 12
Participants
  Baseline | 5 | 3 | 3 | 2 | 2
  Day 6 | 8 | 13 | 12 | 10 | 11

14. Secondary Outcome: Change From Baseline in Urinary Urgency Questionnaire (Questions 2 to 5 and Questions 7 to 14) at Day 6.
Description: Question 2 to Question 6 were assigned scores of 0 to 4 with higher scores indicating worse cases in experience of urinary urgency. Scores for Question 2 to Question 5 were pooled, with a maximum possible score of 16.
  Question 6 was excluded from the analysis since it was only asked at screening. Question 7 to Question 14 were also assigned scores of 0 to 4 with higher scores indicating worse cases in impact of urinary urgency on life; scores for these questions were pooled, with a maximum possible score of 32.
  Baseline was defined as last pre-dose evaluation; Day 6 was defined as Day 6 of Period 1, Day 13 of Period 2 and Day 20 of Period 3.
Time Frame: Day 6
Population: All participants who had taken study drug and have measurements of the pharmacodynamic endpoint were included.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | MR 20 mg | MR 20+20 mg | MR 60 mg | MR 120 mg | IR 90+30 mg
Number analyzed (Participants) | 17 | 17 | 17 | 12 | 12
Units on a scale
  Urinary urgency questionnaire-Question (Q) 2 to Q5 | 1.4 (2.1) | 3.2 (2.4) | 3.2 (3.1) | 4.6 (3.9) | 4.7 (3.0)
  Urinary urgency questionnaire-Q 7 to Q 14 | 0.9 (1.2) | 4.2 (5.5) | 3.5 (5.0) | 10.9 (10.9) | 8.8 (9.8)

15. Secondary Outcome: Number of Participants Experiencing Urinary Frequency Based on Urinary Frequency Questionnaire (Question 1) at Baseline and Day 6.
Description: The ADPKD Urinary Frequency Questionnaire: Question 1 (currently experiencing frequency) was assigned 'Yes' or 'No' to measure current urine frequency status.
  Baseline was defined as last pre-dose evaluation; Day 6 was defined as Day 6 of Period 1, Day 13 of Period 2 and Day 20 of Period 3.
Time Frame: Baseline and Day 6
Population: All participants who had taken study drug and have measurements of the pharmacodynamic endpoint were included.
Measure: Number; unit: Participants
Arm/Group | MR 20 mg | MR 20+20 mg | MR 60 mg | MR 120 mg | IR 90+30 mg
Number analyzed (Participants) | 17 | 17 | 17 | 12 | 12
Participants
  Baseline | 5 | 4 | 4 | 4 | 4
  Day 6 | 10 | 15 | 16 | 12 | 12

16. Secondary Outcome: Change From Baseline in Urinary Frequency Questionnaire (Question 2 and Questions 3 to 10) at Day 6.
Description: Question 2 asked, "During the last 5 days, how much has urinary frequency bothered you?" In order to score the response, the written answers were assigned values from 0 to 4 as follows: 0) Not at all, 1) Somewhat, 2) Moderately, 3) Quite a bit, and 4) Constantly.
  Question 3 to Question 10 were assigned scores of 0 to 4 with higher scores indicating worse cases in impact of urinary frequency on life; scores for these questions were pooled, with a maximum possible score of 32.
  Baseline was defined as last pre-dose evaluation; Day 6 was defined as Day 6 of Period 1, Day 13 of Period 2 and Day 20 of Period 3.
Time Frame: Day 6
Population: All participants who had taken study drug and have measurements of the pharmacodynamic endpoint were included.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | MR 20 mg | MR 20+20 mg | MR 60 mg | MR 120 mg | IR 90+30 mg
Number analyzed (Participants) | 17 | 17 | 17 | 12 | 12
Units on a scale
  Urinary frequency questionnaire-Question (Q) 2 | 0.4 (0.6) | 1.1 (1.1) | 0.9 (0.9) | 1.7 (1.4) | 1.5 (1.1)
  Urinary frequency questionnaire-Q 3 to Q 10 | 1.4 (2.1) | 4.6 (6.9) | 4.1 (5.7) | 12.2 (11.0) | 9.1 (10.5)

17. Secondary Outcome: Ranking of Treatment Tolerability.
Description: Ranking of treatment tolerability was evaluated based on a questionnaire. At Day 22, participants were asked the following questions and their responses recorded on the eCRF: "Which treatment period did you find most tolerable?" and "Which treatment period did you find the least tolerable?".
Time Frame: Day 22/Early Termination
Population: All participants who had taken study drug and have measurements of the pharmacodynamic endpoint were included.
Measure: Number; unit: Participants
Arm/Group | MR 20 mg | MR 20+20 mg | MR 60 mg | MR 120 mg | IR 90+30 mg
Number analyzed (Participants) | 17 | 17 | 17 | 12 | 12
Participants
  Most tolerable Group 1: number analyzed (Participants) | 4 | 4 | 4 | 12 | 12
  Most tolerable Group 1 | 3 | 2 | 3 | 1 | 1
  Most tolerable Group 2: number analyzed (Participants) | 13 | 0 | 13 | 0 | 0
  Most tolerable Group 2 | 10 |  | 3 |  |
  Least tolerable Group 1: number analyzed (Participants) | 4 | 0 | 0 | 12 | 12
  Least tolerable Group 1 | 0 |  |  | 4 | 6
  Least tolerable Group 2: number analyzed (Participants) | 13 | 13 | 13 | 0 | 0
  Least tolerable Group 2 | 0 | 7 | 6 |  |

ADVERSE EVENTS:
Time Frame: Screening to seven days (+ 1 day) after the last dose of study medication.
Description: In safety analysis, all participants who had taken at least one dose of study medication were included.
Arm/Group | MR 20 mg | MR 20+20 mg | MR 60 mg | MR 120 mg | IR 90+30 mg
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/17 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 5/17 | 10/17 | 6/17 | 8/12 | 7/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MR 20 mg (N=17) | MR 20+20 mg (N=17) | MR 60 mg (N=17) | MR 120 mg (N=12) | IR 90+30 mg (N=12)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0
Feeling cold (General disorders) | 1 | 0 | 0 | 1 | 0
Feeling hot (General disorders) | 1 | 0 | 1 | 0 | 0
Mucosal dryness (General disorders) | 0 | 0 | 0 | 1 | 0
Thirst (General disorders) | 1 | 3 | 2 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Polydipsia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 2 | 3
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 2 | 1 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Nervousness (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 2 | 2 | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 1 | 2 | 1 | 1 | 3
Pollakiuria (Renal and urinary disorders) | 2 | 2 | 1 | 2 | 0
Polyuria (Renal and urinary disorders) | 2 | 5 | 1 | 4 | 5
Renal pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No